CLINICAL TRIAL: NCT06488183
Title: Laparoscopic Preperitoneal Local Anesthetic Infiltration Versus Ultrasound Guided Quadratus Lumborum Block in Laparoscopic Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: sarah mohamed (Other)
Responsible Party: Sponsor-Investigator, sarah mohamed, MD, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0306673
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Pain Management
Keywords: preperitoneal infiltration , bariatric surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group p (Other): laparoscopic preperitoneal local anesthetic infiltration
  Interventions: Procedure: preperitoneal local anesthetic infiltration in group p , quadratus lamborum block in group Q
- group Q (Other): ultrasound guided quadratus lamborum block
  Interventions: Procedure: preperitoneal local anesthetic infiltration in group p , quadratus lamborum block in group Q

INTERVENTIONS:
Procedure: preperitoneal local anesthetic infiltration in group p , quadratus lamborum block in group Q — preperitoneal local anesthetic infiltration in group p quadratus lamborum block in group Q

SUMMARY:
preperitoneal local anesthetic infiltration is effective for relief of postoperative pain in patients undergoing laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
Obesity and overweight have become a global epidemic, impacting people of all ages and socioeconomic status. Obesity is still a major public health issue globally, despite progress in some places. Bariatric surgery remains the most effective and long-lasting way to lose weight and address obesity-related conditions.(1) Optimizing postoperative pain treatment is crucial for reducing complications, shortening hospital stays, and lowering expenditures in patients undergoing surgery. Multimodal analgesia and postoperative pain reduction are especially relevant to bariatric surgery patients, who frequently have numerous coexisting conditions and are more vulnerable to thrombotic and respiratory problems. Obstructive sleep apnea (OSA) is common among obese individuals, making safe analgesic treatment problematic. Controlling pain following bariatric surgery is particularly difficult. General management recommendations include multimodal analgesic therapy, regional methods, avoidance of sedatives and early mobilization.(2, 3, 4, 5)

Blanco originally described the quadratus lumborum block (QLB) in 2007. The primary benefit of QLB is the extension of a local anesthetic agent beyond the transversus abdominis plane into the thoracic paravertebral area. The greater distribution of local anesthetic agents may provide significant analgesia and prolong the action of the injected local anesthetic solution.(6)

Preperitoneal local anesthetic injection was initially developed by Dean et al. as a pain management strategy for laparoscopic hernia repair, and it is currently widely used.(7) A recent meta-analysis compared preperitoneal and subcutaneous wound catheters to epidural analgesia. Preperitoneal wound catheters were shown to be as effective as epidural analgesia in abdominal surgeries. Periportal wound catheters appear to be more effective in terms of patient satisfaction and recovery.(8) A recent study concluded that preperitoneal local anesthetic infiltration is effective for relief of postoperative pain in patients undergoing laparoscopic bariatric surgery.(9)

Aim of the work:

The present study aims to compare the analgesic efficacy of ultrasound-guided trans-muscular quadratus lumborum block (QLB) to preperitoneal local anesthetic infiltration during laparoscopic bariatric surgery and in the early postoperative period.

Primary outcome:

• Postoperative pain score

Secondary outcomes:

* Intraoperative fentanyl requirements
* Postoperative morphine requirements
* Time to first dose of rescue analgesia
* Postoperative nausea and vomiting
* Length of stay in PACU
* Early mobilization
* Length of hospital stay

Patients :

Study settings:

This study will be conducted in general surgery department, Alexandria university hospitals.

Study design:

Double blind, randomized, prospective and controlled study

Sample size calculation:

Based on previous study(10, 11), we would need a minimum sample size of 44 participants (22 in each group) to reliably detect an effect size of δ≥ 0.883, assuming a two-sided criterion for detection that allows for a maximum type I error rate of a= 0.05 that achieve 80% power.

Table 1 - Sample Size and Power Analysis User Defined Group P LPLAI Group Q QLB Effect Size Power α 22 22 0.883 0.800 0.0500

The power analysis of sample size (22) in this study equals 0.80, this indicates there is an 80% probability that the statistical test used in our study will correctly reject the null hypothesis.

Study population:

All patients will be randomized 1:1 using a sealed envelope method. Patients will be divided into two equal groups:

Group Q: patients will undergo laparoscopic bariatric surgery under general anesthesia and bilateral ultrasound guided quadratus lamborum block (QLB).

Group P: patients will undergo laparoscopic bariatric surgery under general anesthesia and preincisional laparoscopic preperitoneal bupivacaine infiltration.

Inclusion criteria:

1. Age: 20-50 years, both sexes.
2. ASA physical status class I to III.
3. BMI 35-50 kg/m²

Exclusion criteria:

1. Severe cardiac disorder
2. chronic renal failure
3. liver cirrhosis
4. allergy to bupivacaine
5. patients with history of chronic opioid consumption
6. HBA1C > 7%

Methods:

Preoperative evaluation and preparation:

During preoperative visit, evaluation of patients will be carried out through proper history taking, clinical examination and routine laboratory investigations including complete blood picture, coagulation profile, blood urea, serum creatinine, serum electrolytes, fasting blood glucose, glycosylated haemoglobin (HBA1C), liver function tests and any other investigation needed.

Pre-anesthetic preparation and premedication:

* Informed written consent, from all individual participants who will be included in this study will be taken during preoperative visit.
* Patients should be trained during preoperative visit on a visual analogue scale (VAS), with 0 corresponding to no pain and 10 to the worst pain imaginable.
* Patients will be informed about the analgesic regimen
* Thrombotic prophylaxis (enoxaparin 40 mg) will be started 12 hours before surgery.

On arrival to operative theatre, intravenous cannula will be inserted and standard monitoring will be established using multichannel monitor (Carescape Monitor B650, GE Healthcare Finland) to monitor the following in both groups:

* Electrocardiogram (ECG) for heart rate and rhythm. (Beats/min).
* Non-invasive measurement of arterial blood pressure. (Mean blood pressure in mmHg).
* Pulse oxygen saturation. (SpO2%).
* End tidal CO2 tension (in mmHg).
* Entropy

Anesthesia:

After preoxygenation for 3 minutes, anesthesia will be induced in both groups with propofol 2mg/kg of lean body weight until loss of verbal response, fentanyl 2µg/kg and atracurium 0.5 mg/kg intravenously. Anesthesia will be maintained by isoflurane with 50% oxygen in air (1.2-1.5 %) to maintain entropy between 40-60. Mechanical ventilation will be performed with tidal volume of 8 ml/ kg and a respiratory rate of 12-15 cycles/min to maintain the end-tidal carbon dioxide tension between 35 and 40 mmHg and an oxygen saturation of ≥ 98 per cent with 50 percent oxygen in air. Incremental doses of atracurium will be given every 30 minutes to maintain muscle relaxation. In both groups, signs of insufficient analgesia (eg, tachycardia over 20% of the preoperative value occur during anesthesia) or somatic response (eg, movement ,tearing ,or sweating), will be treated with additional boluses of fentanyl 0.5 mcg/kg intraoperatively as needed. Intraoperatively, all patients will receive IV dexamethasone (8 mg), paracetamol (1 g), ketorolac (30 mg).

All patients in group Q will receive bilateral injection of 30ml bupivicaine 0.25% between quadratus lumborum and psoas major muscles after induction of general anesthesia. Patients in group P will receive 60 ml bupivacaine 0.25% in the preperitoneal space from all quadrants around each trocar and will be held in trendeleberg's position for 5 minutes.

Technique of ultrasound guided quadradus lumborum block:(12) The patient will be placed in the lateral position with the side to be anesthetized turned upwards. Skin preparation with povidone iodine solution will be done, and curvilinear transducer will be placed in the transverse plane at the abdominal flank immediately cranial to the iliac crest. Then the transducer will be moved dorsally keeping the transverse orientation until the quadratus lumborum muscle will be identified with its attachment to the lateral edge of the transverse process of the L4 vertebral body. The needle will be inserted in-plane to the transducer and advanced till penetrating the ventral proper fascia of the quadratus lumborum muscle and 30 ml bupivacaine 0.25% will be injected between the quadratus lumborum and psoas major. The procedure will be repeated on the opposite side.

Technique of laparoscopic preperitoneal local anesthetic infiltration:(10) The patient will be placed in the supine position on the bed with both arms secured to the footboard. Pneumoperitoneum will be achieved via a Veress needle at the Palmer's point. A camera incision will be made 16 cm from the xiphoid process and 1 cm to the left midline. An 11mm port trocar was inserted; a 5mm camera size will be used to explore the abdomen. With the guidance of the camera, the second skin incision will be made for 15mm port, 1 cm proximal, and 5 cm to the right of the first incision. The third incision (5mm) will be made 1 cm proximal and 5 cm to the left side of the patient. The fourth incision (5mm) will be made 1 - 3 cm to the left of the xiphoid process. After skin incisions were made, a Veress needle will be inserted until it reach the preperitoneal space under laparoscopic guidelines with infiltration of 60 ml of bupivacaine 0.25% . The periperitoneum space will be infiltrated adequately from all the quadrants around each trocar. Only the camera port will be infiltrated after the trocar placement. The infiltration takes 20 - 30 seconds for each port.

At the end of surgery, awake extubation, in a semi-sitting position, will be done. Then, the patient will be transferred to the PACU. In PACU, all patients will be assessed for presence and severity of pain; using Visual Analog Scale (VAS). Patients will be prescribed IV morphine 0.1 mg/kg of lean body weight boluses on 4-6 hours basis with a maximum of 10 mg if VAS > 3. Pain control in the ward will be achieved with IV paracetamol 1 g every 6 hours and ketorolac 30 mg every 12 hours. Outcome assessors in PACU and ward will be blinded to patient group assignment and to the nature of the study.

Measurements:

The following data will be measured:

I- Demographic data:

Patient's age (years), sex, body mass index (BMI) (kg/m2 ) and co-morbidities will be recorded.

II- Haemodynamic measurements:

* Pulse rate (Beat / min).
* Non-invasive measurement of mean arterial blood pressure (in mmHg)
* Pulse oxygen saturation All previous parameters will be continuously monitored and recorded before induction of anesthesia, after anesthesia and every 30 minutes until end of surgery.

III- Intraoperative fentanyl requirements (mcg). IV- length of stay in PACU (minutes). V- Assessment of pain using VAS at 1, 2, 4, 6, 12 and 24 hours postoperatively. VI- Time to first morphine dose. VII- Postoperative morphine requirements (mg) VIII- Postoperative nausea and vomiting IX- length of hospital stay (days).

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-50 years, both sexes.
* ASA physical status class I to III.
* BMI 35-50 kg/m²

Exclusion Criteria:

* Severe cardiac disorder
* chronic renal failure
* liver cirrhosis
* allergy to bupivacaine
* patients with history of chronic opioid consumption
* HBA1C > 7%

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | postoperative day 1
  VAS score

SECONDARY OUTCOMES:
postoperative morphine requirements | postoperative day 1
  mg
postoperative nausea and vomiting | postoperative day1
  number
length of stay in pacu | postoperative day 1
  minutes
Length of hospital stay | postoperative day 3
  days

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aldohayan A, Alshammari S, Binjaloud A, Bamehriz F, Narejo AS, Aqil M, Aldahian N, Aldabaeab A, Eldawlatly A. Pre-incisional Laparoscopic Preperitoneal Local Anesthetic Technique in Laparoscopic Sleeve Gastrectomy. JSLS. 2022 Jul-Sep;26(3):e2022.00049. doi: 10.4293/JSLS.2022.00049. PMID 36071990